CLINICAL TRIAL: NCT02356367
Title: French Cohort Study of Chronic Heart Failure Patients With Central Sleep Apnoea Eligible for Adaptive Servo-Ventilation (PaceWave, AutoSet CS, AirCurve 10 CS): Predictive Factors of Poor Compliance
Brief Title: French Cohort Study of Chronic Heart Failure Patients With Central Sleep Apnoea Eligible for Adaptive Servo-Ventilation (PaceWave, AutoSet CS, AirCurve 10CS): Predictive Factors of Poor Compliance (FACE)
Acronym: FACE
Status: Withdrawn | Type: Observational
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Other Study IDs: Face Pilot Study
Record Dates: First submitted 2015-02-02; First posted 2015-02-05 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Central Sleep Apnea; Heart Failure
Keywords: telemonitoring; Adaptive servo-ventilation
MeSH Terms: conditions — Sleep Apnea, Central; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: telemonitoring
  Other Names: Airview

SUMMARY:
The purpose of this study is to determine the predictive factors of poor compliance to sleep disordered breathing therapy in chronic heart failure patients treated for central sleep apnea. To characterize nocturia pathophysiology associated with SDB in this population. To use telemonitoring data to define predictive factors of poor compliance.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patient with Chronic Heart Failure
* Central Sleep Apnea requiring Adaptative Servo-Ventilation therapy
* Patient is able to fully understand study information and signed informed consent

Exclusion Criteria:

* Contra-indications to Adaptative Servo-Ventilation therapy
* Respiratory Failure or Hypercapnia inconsistent with Adaptative Servo-Ventilation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart Failure patient eligible for adaptative servo-ventilation
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
to define the phenotype of compliant or not compliant patients to sleep disordered breathing therapy using microneurography | 12 months
  Autonomic nervous system balance measure by microneurography

SECONDARY OUTCOMES:
anxiety and nervous depression | 12 months
  using Spielberger questionnaire and Beck's Depression Inventory
sleep disordered breathing symptomatology | 12 months
  using Epworth sleepiness scale and Oxford Sleep Resistance Test
Nocturia | 24 months
  evaluated by number of urination per night, diuresis, plasmatic dosage of Atrial Natriuretic peptide, Brain natriuretic peptide, Antidiuretic hormone
sleep quality | 24 months
  evaluated by Pittsburgh Sleep Quality Index; minnesota living with heart failure questionnaire; actimetry; home polysomnography
Heart Failure status | 24 months
  evaluated by echocardiography, New York Heart Association functional classification; Electrocardiography
therapy compliance | 24 months
  evaluated by Morisky Medication Adherence Scale and with telemonitoring data

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU Henri Mondor, Créteil
  - CHU de Grenoble, Grenoble
  - CHU Bichat, Paris